CLINICAL TRIAL: NCT03862183
Title: Survey on BP, Lipids and Cardiovascular Risks in the Outpatient Hypertensives and Continuing Medical Education Program
Brief Title: Hospital-level Variation in the Management of Blood Pressure and Low-density Lipoprotein in the Outpatient Hypertensives in China-a Cross Sectional Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Huashan Hospital (Other)
Responsible Party: Principal Investigator, Yong Li, associate chief of the cardiology department, Huashan Hospital
Other Study IDs: UPPDATE
Record Dates: First submitted 2019-03-02; First posted 2019-03-05 (Actual); Last update posted 2019-03-05 (Actual); Status verified 2019-03

CONDITIONS: Hypertension; Hyperlipidemia
MeSH Terms: conditions — Hypertension; Hyperlipidemias

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- dyslipidemia in hypertension
  Interventions: Other: continuing medical education program
- hypertension
  Interventions: Other: continuing medical education program

INTERVENTIONS:
Other: continuing medical education program — educating all the involved doctor the same medical knowledge on hypertension control

SUMMARY:
To investigate the proportion, medication use and control rate of metabolic abnormalities such as dyslipidemia in outpatients with hypertension in different levels of hospitals in China. To investigate the gap between guidelines and clinical practices, and analyze the cause. we also set up a continuing medical education program to narrow the gap and the effect of the program will be estimated.

ELIGIBILITY:
Inclusion Criteria:

1. Outpatients from departments of Cardiology, Endocrinology, Nephrology, Neurology, Geriatrics or General Internal Medicine.
2. Diagnosed as hypertension. Diagnostic criteria: 1)The office BP measured at the day of visit and at least one time before that day were above the cut-off values ( ≥140 mmHg SBP and/or ≥90 mmHg DBP); 2)for patients with normal BP at the day of visit, they should have already been given pre-treatment with antihypertensive drugs ≥ 2 weeks.
3. Voluntary participation.

Exclusion Criteria:

1. Patients aged< 18 years old.
2. Patients without a definite diagnosis of hypertension（for instance, if the patient has been taking antihypertensive drugs irregularly, it is difficult to confirm the diagnosis of hypertension）.
3. Patients with a definite diagnosis of secondary hypertension.
4. Patients are diagnosed dyslipidemia with clear cause, such as nephrotic syndrome, severe hypothyroidism, terminal stage of malignancy, etc.
5. Patients are diagnosed end-stage renal disease, hemodialysis, and peritoneal dialysis patients.
6. Patients diagnosed with mental abnormalities who are unable to complete the questionnaire.
7. Patients have once participated in this research during this study cycle（to avoid repeated participation）.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: outpatients with hypertension in different levels of hospitals in China
Sampling Method: Non-Probability Sample
Enrollment: 21000 (Estimated)
Dates: Start 2017-07-01 (Actual); Primary Completion 2020-12-30 (Estimated); Study Completion 2020-12-30 (Estimated)

PRIMARY OUTCOMES:
rate of blood pressure goal achievement | 2017-2020
  systolic blood pressure<140mmHg and diastolic blood pressure<90mmHg

CONTACTS AND LOCATIONS:
Locations (1):
- Cardiology Department in Huashan Hospital, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Derived] Xie K, Gao X, Bao L, Shan Y, Shi H, Li Y. The different risk factors for isolated diastolic hypertension and isolated systolic hypertension: a national survey. BMC Public Health. 2021 Sep 14;21(1):1672. doi: 10.1186/s12889-021-11686-9. PMID 34521364